CLINICAL TRIAL: NCT06287801
Title: Supporting Practices In Respecting Elders Phase 1
Brief Title: Annual Wellness Visits vs GRACE-augmented Annual Wellness Visits For Older Adults With High Needs - Phase 1
Acronym: SPIRE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brandeis University (Other); Vanderbilt University Medical Center (Other); Dartmouth-Hitchcock Medical Center (Other); Indiana University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Christine S. Ritchie, MD, MPH, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024P000271
Record Dates: First submitted 2024-02-13; First posted 2024-03-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging; Health Care Utilization; Health-Related Behavior
Keywords: high-risk elderly; ACO; Medicare; Annual Wellness Visits (AWV); Geriatric collaborative care
MeSH Terms: conditions — Patient Acceptance of Health Care; Health Behavior | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Feasibility of a clinical comparative effectiveness trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor team will be blinded to the intervention assignments of participants. Due to the nature of the intervention, the participants, the investigator, and the care providers are unable to be blinded to the participant assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Annual Wellness Visits (AWV) (Experimental): Randomized Vanderbilt Health Affiliated Network (VHAN) practice to AWV and assess impact on the population deemed by study algorithm as high-risk and recruit 50 participants from the VHAN primary care clinical practice (n=50/practice) to complete surveys prior to the intervention and 6 months later.
  Interventions: Other: Annual Wellness Visit
- Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE) (Experimental): Randomized Vanderbilt Health Affiliated Network (VHAN) practice to AWV + GRACE and assess impact on the population deemed by study algorithm as high-risk and recruit 50 participants from the VHAN primary care clinical practice (n=50/practice) to complete surveys prior to the intervention and 6 months later.
  Interventions: Other: Annual Wellness Visit; Other: Geriatric Resources and Assessment for the Care of Elders

INTERVENTIONS:
Other: Annual Wellness Visit — Completion of a structured Annual Wellness Visit (AWV) questionnaire administered by an assigned practice staff member for Medicare beneficiaries deemed by study algorithm as high-risk. Those responses will then be used by the primary care team to place any needed referrals and offer any indicated personal health advice and create a care plan for the coming year. Routine usual care from the primary care practice will occur.
  Other Names: AWV
Other: Geriatric Resources and Assessment for the Care of Elders — The practice will initiate the Geriatric Resources and Assessment for the Care of Elders (GRACE) program for Medicare beneficiaries deemed by study algorithm as high-risk and meeting other study criteria (see below). After completion of the in-home structured annual wellness visit (AWV) and GRACE assessment by the NP/SW team, responses will be reviewed and applied to construct an individualized care plan using the GRACE protocols inclusive of advance care planning, health maintenance, medication management, assistance with any difficulty walking, falls, dementia, depression, chronic pain, malnutrition, weight loss, urinary incontinence, visual impairment, hearing impairment, or caregiver burden.
  Other Names: GRACE
  Arms: Annual Wellness Visits + Geriatric Resources and Assessment for the Care of Elders (AWV + GRACE)

SUMMARY:
This study consists of three aims focused on examining the feasibility of adding the Geriatric Resources and Assessment for the Care of Elders (GRACE) model to structured Annual Wellness Visits (AWVs) to improve patient and caregiver outcomes and reduce hospitalizations in older adults with complex health needs. The objectives are to:

1. Co-design a community-centric implementation strategy for the AWVs vs AWVs + GRACE -augmented care (AWV GRACE) study arms
2. Develop a referral pathway and algorithm to optimize enrollment of eligible participants
3. Conduct a pilot clinical trial to assess the feasibility of the AWV GRACE intervention.

DETAILED DESCRIPTION:
In the United States, 10% of patients account for half of health care costs. Many of these are older adults with complex health and social care needs (referred to as "older adults with complex needs"). They see a doctor on average 9.6 times per year, 3 times more often than older adults overall. Patients, caregivers/care partners experience care as confusing and disorganized (the investigators will refer to caregivers and care partners interchangeably here, reflecting preferences of our stakeholder reviewers). Clinicians in primary care practices and accountable care organization leaders (ACOs) face critical dilemmas about how best to care for older adults with complex needs. Patient stakeholders providing feedback on preferred care models worry about fragmented care. Many also prefer to be at home.

Evidence suggests that optimal care of older adults with complex needs involves an interprofessional team of doctors, nurses, social workers and other health care staff in partnership with patients and care partners to provide person-centered care plans, guided by evidence-based geriatric assessments. Few primary care practices provide this type of care, but Medicare ACOs and other value-based care models such as Medicare Advantage plans are well positioned to link clinicians and provide support for complex patients, their caregivers and care partners. ACOs are groups of clinicians, often housed in healthcare systems, who share in savings if they deliver high-quality care. Unlike traditional fee-for-service payment arrangements, the payment models in ACOs reward efficient, patient centered care that also minimizes unhelpful (and sometimes harmful) institutional care. ACOs are eager to optimize effective care for their patients with complex needs, but best strategies are unknown. ACO stakeholders working with us in the development of this proposal seek effective approaches to care for their older adult patients with complex needs and report readiness to engage in collaborative processes to develop alternate care models. Medicare Advantage (or Medicare Part C) is a capitated form of value based care, which is rapidly growing in market share among Medicare beneficiaries.

In 2011, Annual Wellness Visits (AWVs) were introduced as a Medicare Part B benefit on January 1st 2011. AWVs seek to incorporate routine geriatric assessments in primary care practices of older adults' to produce a Personalized Preventive Plan (PPP) to be reviewed with the patient by primary care clinical staff. AWVs have required elements which need to be addressed by a health provider, who then files charges to CMS for the administration of these services. However, there is wide variation in the approach to administration of the AWV (ranging from in-person interviews by physician and non-physician practitioners to completion by the patient or caregiver prior to the visit using self-report questionnaires. While uptake by clinicians has accelerated, uptake is lower for more older adults who face disparities in care due to income, race and ethnicity. In Medicare Shared Savings Program (MSSP) ACOs, 55% of beneficiaries received an AWV in 2021. Yet among adults 75-85 years old who were dually eligible for Medicaid and Medicare, fewer than half (42%) received an AWV (authors' analysis of Institute for Accountable Care Medicare Part B claims). In addition, office-based AWV's are not necessarily oriented to high-need, complex older adults, who warrant more nuanced attention to their living environment and longitudinal care needs. Few interventions have pursued the study of a more robust AWV conducted in patients' homes and linked to clear geriatric care paths in an effort to more effectively navigate the biopsychosocial needs of this aging population.

The Geriatric Resources and Assessment for the Care of Elders (GRACE) Program offers an evidence-based approach to support geriatric assessment and care planning for complex patients receiving AWVs. GRACE is a protocolized interprofessional co-management model that was developed to improve the patient experience of care, provide patients and caregivers with a designated point of contact, reduce utilization costs, and support overburdened primary care providers by co-managing complex patients. The care plan was built collaboratively (including patients and family caregivers) using GRACE Protocols for common geriatric conditions and provides a checklist to ensure a standardized approach to care. GRACE protocols were also developed in partnership with primary care physicians and address 12 common geriatric conditions to support and complement primary care: advance care planning, health maintenance, medication management, difficulty walking/falls, malnutrition/weight loss, visual impairment, hearing loss, dementia, chronic pain, urinary incontinence, depression, caregiver burden. Even though GRACE has been demonstrated in a randomized controlled trial among patients at high risk for hospital to improve quality and decrease cost, GRACE has not been adopted by the majority of ACOs, in contrast to the more common use of AWVs.

Based on our hypothesis that patients with complex needs require annual wellness visits and an integrated program of complex care management (i.e., AWVs + GRACE) to achieve improved health outcomes and a commitment from our proposed study partners to fund additional staff to support AWV + GRACE care delivery, the investigators plan to study the intervention AWVs + GRACE as defined by the following components:

1. The investigators will apply a community-engaged approach and co-design an optimal implementation strategy for effectively delivering structured AWVs vs. AWVs with GRACE-augmented care (AWV GRACE). Stakeholder input from Vanderbilt Health Affiliated Network (VHAN) clinical teams, clinical and community leads and other health system collaborators will inform the formation and operation of implementation support communities, implementation coaching, and technical assistance. This process will guide specific adaptations of these implementation domains for high-need older adults within accountable care organization (ACO) and Medicare Advantage- supported primary care practices.
2. The investigators will assess existing ACO algorithms for identifying older adults with complex needs and determine which criteria are most appropriate for inclusion in the study for screening and enrollment at two primary care practices within the VHAN for a pilot trial to be performed (discussed below). Based on input from our stakeholder working groups, the investigators will build statistical models and referral pathways to more accurately identify high need older adult populations and refine our eligible populations and confirm our sample size requirements.
3. The investigators will determine the feasibility of conducting a clinical comparative effectiveness trial of structured AWV alone vs. AWV + GRACE at two primary care practices within Vanderbilt Health Affiliated Network (VHAN) by conducting a pilot trial. Designated VHAN primary care practices (N=2) will be randomized to the intervention (AWV GRACE) or the control arm (AWV) and practice staff will be trained to deliver the assigned intervention per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. be 65 years of age or older
2. be eligible for an AWV during the study period
3. have a residential mailing address within a 45-mile radius of the Vanderbilt clinics
4. have a working home/mobile telephone number where they can be reached
5. be English or Spanish speaking
6. be able to provide consent and /or have a proxy able to consent to study participation

Exclusion Criteria:

1. are receiving hospice care
2. are currently housed at Long Term Care Facilities
3. are incarcerated

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Hospitalizations | Up to 12 months prior to intervention vs 6 months after intervention
  Rate of inpatient hospitalizations evaluated at the participant level
Consumer Assessment of Healthcare Providers and Systems Clinician and Group Survey (CG-CAHPS) with Patient Centered Medical Home 1.0 supplement (PCMH CAHPS) | Within 1 month of intervention and 6 months after intervention
  The CAHPS Clinician & Group Survey (CG-CAHPS) asks patients to report on their experiences with providers and staff in primary care and specialty care settings, using a 6 month recall period. The Patient-Centered Medical Home (PCMH) Item Set is a set of supplemental questions that is added to the adult version of the CAHPS Clinician & Group Survey (CG-CAHPS) to gather more information on patient experience with the domains of primary care that define a medical home.
  Scoring for most items is on a 4 point scale 1=never 2=sometimes 3=usually 4=Always. Minimum and Maximum scores vary with the number of items used. The Provider Rating item is on a 11 point scale from 0 to 10,where 9,10 are considered "high" scores.
Net Promotor Score | Within 1 month of intervention and 6 months after intervention
  The single question - "How likely are you to recommend X to a friend [or colleague]?" is rated from 0 - Not at all likely to 10 - Extremely likely.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health - Physical Health (PH) and Mental Health (MH) | Within 1 month of intervention and 6 months after intervention
  These measures are derived from 10 items covering self-reported assessment of physical health, physical functioning, pain intensity, fatigue, overall quality of life, mental health, satisfaction with social activities, and emotional problems. Items are scored on a 1-5 Likert scale.
Caregiver Strain | Within 1 month of intervention and 6 months after intervention
  We will use the Modified Caregiver Strain Questionnaire-Short Form developed originally by Bickman and revalidated for use with caregivers of older adults to assess the subjective and objective burden of care-giving. The tool asks about events (financial stress) or feelings (guilt) as a result of caring for a family member with chronic health problems.
  There are 13 items, each item is scored from 0 to 2 (0=no, 1=yes, sometimes, and 2=yes, on a regular basis), and total scores can range from 0 to 26. Any positive response may indicate a need for intervention in that area. Higher scores on the MCSI indicate greater caregiver strain; a score of 7 or higher indicates a high level of stress
Patient's out-of-pocket costs for up to 180 days after enrollment | Up to 6 months after enrollment
  Within Medicare, out-of-pocket costs can vary depending on things like the length of an inpatient stay or the choice to administer a drug at home versus in the hospital. As a result, we will assess patient out of pocket costs for the two study arms using Medicare claims data. These data include details on all copayment and deductible paid by Medicare beneficiaries.
Caregiver's hours spent caregiving. | Within 1 month of intervention and 6 months after intervention
  As care shifts from institutional to home and community-based settings, one potential unintended consequence is increased caregiver burden. Although we are already assessing caregiver strain, a measure of psychological distress, we will add a focused assessment of the amount of time dedicated to caregiving. These data will be collected via survey
Pilot ACOs Staffing costs | At the completion of the pilot phase
  To assess this, we will ask each participating ACO to complete an annual costing worksheet that has been developed by the Institute for Accountable Care as part of a return-on-investment tool commonly shared with ACOs.

OTHER OUTCOMES:
Exploratory Geriatric Outcomes - Number of participants with new ICD-10 diagnosis codes | Within 1 month of intervention and 6 months after intervention
  New ICD-10 diagnosis codes in cognitive status, physical function status or mood categories
Exploratory Geriatric Outcomes- number of participants that complete advanced care planning documents | Within 1 month of intervention and 6 months after intervention
  Completion of health care proxy or advance care planning documents
Exploratory Geriatric Outcomes - number of participants with inappropriate medications | Within 1 month of intervention and 6 months after intervention
  Numbers of potentially inappropriate medications
Covariate - Demographics | Within 1 month of intervention
  age, sex, race/ethnicity
Covariate - Medicare Entitlement Status | Within 1 month of intervention
  Identify patients as Medicare qualifying due to age, non-dual Medicare, dually eligible for Medicaid and Medicare, disabled Medicare, end-stage renal disease Medicare entitlement status
Covariate - Elixhauser comorbidity index | Within 1 month of intervention and 6 months after intervention
  The Elixhauser index categorizes 30 morbidities based on the International Classification of Diseases (ICD) codes found in administrative data and is associated with resource use and in-hospital mortality. Each comorbidity category is dichotomous. A weighting algorithm was developed, based on the association between comorbidity and death, in order to produce an overall score for the Elixhauser Index.
Covariate - Area Deprivation Index | Within 1 month of intervention
  The ADI is an indicator of structural barriers to health and well-being that uses the Zip+4 code listed for the patient's residence in the Medicare Beneficiary Summary File to link to the census block group with the same Zip+4 area in US Census data. ADI scores are based on Singh's Census indicators weighted by Singh's factor score coefficients for each indicator.
Covariate - Loneliness | Within 1 month of intervention and 6 months after intervention
  The University of California, Los Angeles (UCLA) 3-item loneliness scale assess relational connectedness, social connectedness and self-perceived isolation.
  The scores for each individual question can be added together to give participants a possible range of scores from 3 to 9. Researchers in the past have grouped people who score 3 - 5 as "not lonely" and people with the score 6 - 9 as "lonely".
Exploratory - Hope | Within 1 month of intervention and 6 months after intervention
  The Hearth Hope Index (HHI) measures hope along three dimensions:
  Temporality and future: This dimension assesses the individual's belief in the future and their ability to set and achieve goals.
  Positive readiness and expectancy: This dimension assesses the individual's sense of optimism and their belief in their ability to overcome challenges.
  Interconnectedness: This dimension assesses the individual's sense of connection to others and their belief in the power of relationships.
  The HHI scale has been shown to be a reliable and valid measure of hope. It has been used in a variety of settings, including clinical practice, research, and education.
  The HHI measures various dimensions of hope using a 4-point Likert scale that ranges from 1 (strongly disagree) to 4 (strongly agree) with items #3 and #6 reverse-coded. The scale has one global score that ranges from 12 to 48, as well as single-item scores that range from 1 to 4; higher scores indicate greater hopefulness.
Covariate - Activities of daily living (ADL) | Within 1 month of intervention and 6 months after intervention
  Activities of daily living rated on a scale of INDEPENDENT (1), NEED HELP (2), DEPENDENT (3), CANNOT DO (4).
Exploratory - ED visits | Up to 12 months prior to intervention vs 6 months after intervention
  Rate of emergency department visits that do not result in an inpatient hospitalization evaluated at the participant level
Exploratory - Observation visits | Up to 12 months prior to intervention vs 6 months after intervention
  Rate of observation visits that do not result in an inpatient hospitalization evaluated at the participant level

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The data can be available by request only after academic journal publication. Any formal requests should be sent by external research teams and will be reviewed by the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available upon request after academic journal publication.
Access Criteria: Access criteria will be determined and confirmed by the corresponding author upon review of the formal data request.

REFERENCES:
- [Background] Conwell LJ, Cohen JW. Characteristics of Persons with High Medical Expenditures in the U.S. Civilian Noninstitutionalized Population, 2002. Published online 2002:6.
- [Background] Feder JL. Predictive modeling and team care for high-need patients at HealthCare Partners. Health Aff (Millwood). 2011 Mar;30(3):416-8. doi: 10.1377/hlthaff.2011.0080. No abstract available. PMID 21383355
- [Background] Weiss KB. Managing complexity in chronic care: an overview of the VA state-of-the-art (SOTA) conference. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):374-8. doi: 10.1007/s11606-007-0379-x. PMID 18026804
- [Background] Grant RW, Ashburner JM, Hong CS, Chang Y, Barry MJ, Atlas SJ. Defining patient complexity from the primary care physician's perspective: a cohort study. Ann Intern Med. 2011 Dec 20;155(12):797-804. doi: 10.7326/0003-4819-155-12-201112200-00001. PMID 22184686
- [Background] High-Need, High-Cost Patients: Who Are They and How Do They Use Health Care? | Commonwealth Fund. Accessed September 3, 2019. https://www.commonwealthfund.org/publications/issue-briefs/2016/aug/high-need-high-cost-patients-who-are-they-and-how-do-they-use
- [Background] Shafir A, Garrigues SK, Schenker Y, Leff B, Neil J, Ritchie C. Homebound Patient and Caregiver Perceptions of Quality of Care in Home-Based Primary Care: A Qualitative Study. J Am Geriatr Soc. 2016 Aug;64(8):1622-7. doi: 10.1111/jgs.14244. Epub 2016 Jul 7. PMID 27384919
- [Background] Sayer C. "Time Spent at Home" - A Patient-Defined Outcome. NEJM Catalyst. Published online April 26, 2016. Accessed December 21, 2022. https://catalyst.nejm.org/doi/abs/10.1056/CAT.16.0854
- [Background] McNabney MK, Green AR, Burke M, Le ST, Butler D, Chun AK, Elliott DP, Fulton AT, Hyer K, Setters B, Shega JW. Complexities of care: Common components of models of care in geriatrics. J Am Geriatr Soc. 2022 Jul;70(7):1960-1972. doi: 10.1111/jgs.17811. Epub 2022 Apr 29. PMID 35485287
- [Background] Auerbach DI, Levy DE, Maramaldi P, Dittus RS, Spetz J, Buerhaus PI, Donelan K. Optimal Staffing Models To Care For Frail Older Adults In Primary Care And Geriatrics Practices In The US. Health Aff (Millwood). 2021 Sep;40(9):1368-1376. doi: 10.1377/hlthaff.2021.00401. PMID 34495726
- [Background] Accountable Care Organizations (ACOs) | CMS. Accessed December 19, 2022. https://www.cms.gov/Medicare/Medicare-Fee-for-Service-Payment/ACO
- [Background] Fraze TK, Beidler LB, Briggs ADM, Colla CH. Translating Evidence into Practice: ACOs' Use of Care Plans for Patients with Complex Health Needs. J Gen Intern Med. 2021 Jan;36(1):147-153. doi: 10.1007/s11606-020-06122-4. Epub 2020 Oct 1. PMID 33006083
- [Background] Ochieng N, Damico A, 2023. Medicare Advantage in 2023: Enrollment Update and Key Trends. KFF. Published August 9, 2023. Accessed August 17, 2023. https://www.kff.org/medicare/issue-brief/medicare-advantage-in-2023-enrollment-update-and-key-trends/
- [Background] MLN6775421 - Medicare Wellness Visits. Accessed December 21, 2022. https://www.cms.gov/Outreach-and-Education/Medicare-Learning-Network-MLN/MLNProducts/preventive-services/medicare-wellness-visits.html
- [Background] Huang H, Zhu X, Wehby GL. Primary care physicians' participation in the Medicare shared savings program and preventive services delivery: Evidence from the first 7 years. Health Serv Res. 2022 Oct;57(5):1182-1190. doi: 10.1111/1475-6773.14030. Epub 2022 Jul 18. PMID 35808929
- [Background] Lind KE, Hildreth KL, Perraillon MC. Persistent Disparities in Medicare's Annual Wellness Visit Utilization. Med Care. 2019 Dec;57(12):984-989. doi: 10.1097/MLR.0000000000001229. PMID 31584462
- [Background] Beckman AL, Becerra AZ, Marcus A, DuBard CA, Lynch K, Maxson E, Mostashari F, King J. Medicare Annual Wellness Visit association with healthcare quality and costs. Am J Manag Care. 2019 Mar 1;25(3):e76-e82. PMID 30875175
- [Background] Counsell SR, Callahan CM, Buttar AB, Clark DO, Frank KI. Geriatric Resources for Assessment and Care of Elders (GRACE): a new model of primary care for low-income seniors. J Am Geriatr Soc. 2006 Jul;54(7):1136-41. doi: 10.1111/j.1532-5415.2006.00791.x. PMID 16866688
- [Background] Rodriguez, S, Munevar, D, Delaney, C, Yang, L, Tumlinson, A. Effective Management of High-Risk Medicare Populations. Published online September 2014.
- [Background] Counsell SR, Callahan CM, Tu W, Stump TE, Arling GW. Cost analysis of the Geriatric Resources for Assessment and Care of Elders care management intervention. J Am Geriatr Soc. 2009 Aug;57(8):1420-6. doi: 10.1111/j.1532-5415.2009.02383.x. PMID 19691149
- [Background] Counsell SR, Callahan CM, Clark DO, Tu W, Buttar AB, Stump TE, Ricketts GD. Geriatric care management for low-income seniors: a randomized controlled trial. JAMA. 2007 Dec 12;298(22):2623-33. doi: 10.1001/jama.298.22.2623. PMID 18073358
- [Background] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- [Background] Boult C, Dowd B, McCaffrey D, Boult L, Hernandez R, Krulewitch H. Screening elders for risk of hospital admission. J Am Geriatr Soc. 1993 Aug;41(8):811-7. doi: 10.1111/j.1532-5415.1993.tb06175.x. PMID 8340558
- [Derived] Travison TG, Pham E, Donelan K, Bartels SJ, Carter JA, Corelli K, Counsell SR, Crean M, Flaherty E, Michael C, Moran DS, Murff HJ, Perloff J, Ritchie CS. Assessing the feasibility, acceptability, and efficacy of a pragmatic pilot and full-scale trial to improve care for older adults with complex care needs: The SPIRE study. Contemp Clin Trials. 2025 Dec;159:108072. doi: 10.1016/j.cct.2025.108072. Epub 2025 Sep 2. PMID 40907942